CLINICAL TRIAL: NCT03407560
Title: Use of the Bone Substitute SintLife® in Vertebral Arthrodesis Procedures. A Pilot Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVOD.SintLife
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2018-01

CONDITIONS: Spinal Fusion
Keywords: bone substitute; spinal fusion; lumbar spine disease
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SintLife (Experimental): Use of SintLife putty as bone substitute for spinal fusion in lumbar spine surgery for degenerative diseases.
  Interventions: Device: SintLife

INTERVENTIONS:
Device: SintLife — Patients will be treated for degenerative diseases of the spine, such as lumbar stenosis, spondylolysis and spondylolisthesis, degenerative disc disease.
  The fusion technique used will be the posterolateral arthrodesis of one or more vertebral levels included in the lumbosacral region (L1-S1), obtained by screws and bars, together with a preparation of the transverse processes treated with bone substitute in order to Sintlife obtain new bone formation and then spinal fusion. It is also possible to associate interbody fusion with the use of a cage.

SUMMARY:
This pilot study is to evaluate the potential effectiveness of bone substitute SintLife within the spinal surgery in spinal stabilization applications for degenerative diseases.

In particular, the investigators propose to evaluate:

* the ability of bone regeneration/ fusion, defined as the presence of trabecular bone continuous bridge and absence of radiolucent lines, verified by diagnostic imaging in accordance with the Brantigan scale;
* the patient's state of health, evaluated through the comparison of the functional-symptom pattern between the pre- and post-operative phases, verified by Oswestry Disability Index (ODI), Visual Analogue Scale (VAS) and EuroQol (EQ-5D);
* the safety of the medical device, evaluated through the impact of any adverse events, complications, unexpected reactions, accidents.

STUDY DESIGN This collection of clinical data is set up as pilot study post-marketing. In the study will be included all consecutive patients who require spinal fusion surgery, in accordance with the inclusion and exclusion criteria after signing the informed consent. Patients will be treated and followed postoperatively according to the normal clinical, surgical and therapeutic practice, in place at the Rizzoli Orthopaedic Institute of Bologna.

The total duration of data collection is 36 months:

* the stage of patient enrollment is 18 months from the date of approval of the study by the Ethics Committee of the center;
* the phase of post-operative monitoring is 18 months, with planned at 6, 12 and 18 months follow-up (± 15 days before scheduled date).

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE The vertebral arthrodesis is one of the surgical procedures most used for the treatment of deformities, trauma and degenerative diseases with instability of the spine (Rajaee et al., 2012; Yoshihara and Yoneoka, 2015).

   Using bone grafts and tools, such as metal rods and screws, this procedure creates a fusion between two or more adjacent vertebrae, in order to stabilize the spine.

   The success of fusion, intended as the neo-formation of trabecular bone radiographically detectable, may depend on the characteristics of the bone graft used and its properties as well as the surgical technique used. In the absence of autologous bone the biological process that leads to bone regeneration is characterized by three critical elements: the osteogenic potential, the osteoinductive factors, the osteoconductive scaffold. The ideal bone substitute possesses all three of these properties, combined with excellent compatibility and biological safety (Ludwig et al., 2000; Park et al., 2013).

   The local autologous bone harvested from the iliac crest has been and is still considered the "gold standard" in the treatment of spinal fusion. However, contraindications and potential complications associated with the use of autologous bone are well known (Dimar et al., 2009; Gruskay et al., 2014; Kim et al., 2009; Miyazaki et al., 2009). In order to overcome these limitations, several alternatives have been developed, clinically tested and are today available on the market: growth factors (BMPs) (Carragee et al., 2011; Kannan et al., 2015), allogenic bone or heterologous ( Gupta et al., 2015; Park et al., 2013), demineralized bone matrix (DBM) and synthetic ceramic materials to name a few (Abdullah et al., 2011; Fischer et al., 2013; Hsu et al., 2012) . Despite all of these materials have been extensively studied (Abdullah et al., 2011; Alsaleh et al., 2012; Hsu et al., 2012; Miyazaki et al., 2009) the available data are often uneven in quality, type of study, assessments performed and conclusions reached (Hsu et al., 2012; Kannan et al., 2015; Miyazaki et al., 2009).

   The ceramic bone substitutes of synthetic origin (Nickoli and Hsu, 2014), such as collagen, tricalcium phosphate (TCP) (Dai and Jiang, 2008), calcium phosphate (CaP), calcium sulphate (CaS) and hydroxyapatite (HA), have been designed and developed as osteoconductive scaffolds with characteristics and properties very similar to those of human bone, able to support the regeneration and bone remodeling, and go into slow resorption (Alsaleh et al. , 2012; Gao et al., 2014; Hsu et al., 2012; Kaiser et al., 2014; Kho and Chen, 2008; Korovessis et al., 2005; Lee et al., 2009; Zhou and Lee, 2011) .

   Fin-Ceramica Faenza SpA is a company engaged in the development of innovative solutions in the field of bone regeneration, and one of the latest solutions in the field of bone substitutes proposes the use of hydroxyapatite-based ceramic composites, biomaterials biomimetic new generation (Blackbeard et al., 2013; Zhou and Lee, 2011). Among these biomaterials, SintLife is a bone substitute consisting of Mg-HA crystals nano (sintered at body temperature). pre-clinical and preliminary clinical data show Sintlife the safety of the product and support the ability to use it as a bone substitute for spinal fusion (Brodano Barbanti et al., 2015; Brodano et al., 2014; Manfrini et al., 2013).
2. IDENTIFICATION AND DESCRIPTION OF MEDICAL DEVICE SintLife is an implantable medical device, not active, with bone substitute function.

   SintLife features reabsorbtion cell-mediated. SintLife is a bone substitute, in paste form, consisting of physiological saline (percentage to 46%) and nanocrystals of magnesium-substituted hydroxyapatite (Mg-HA). The Mg2 + ions are introduced within the crystalline cell of HA in the same position and percentage found in the human bone mineral phase. E 'was shown that the presence of Mg2 + deforms the structure of the HAS crystalline cell by making it unstable and biologically active, thus promoting bone formation, remodeling, and a rapid resorption mediated by the cells of the material. In addition, the Mg-HA actively interacts with the water molecules to quickly capture key proteins involved in osteogenesis.

   SintLife interacts with the cells that form bone and promotes the deposition of new bone tissue. Thanks to its specific chemical composition and biomimetics, the nanostructure and the surface properties, it is reabsorbed and remodeled by the action mobile phone in a physiologically appropriate time (6-18 months), remaining at the application site for the duration of growth and of maturation of new bone.

   During the remodeling phase, one can observe the resorbing activity of osteoclasts to work around the particles of the material, until a complete bone regeneration (5). SintLife is classified as a Class III medical device, is CE marked and complies with current European legislation on medical devices (EC Directive 93/42 / EC amended 2007/47 / EC).
3. PURPOSE, OBJECTIVES AND EVALUATION This pilot study is to evaluate the potential effectiveness of bone substitute SintLife within the spinal surgery in spinal stabilization applications for degenerative diseases.

   In particular, the investigators aim to evaluate:
   * the ability of bone regeneration / molding, defined as the presence of trabecular bone continuous bridge and absence of radiolucent lines, verified by diagnostic imaging (CT) and evaluated by means of in accordance with the scale Brantingan
   * the patient's state of health, through the comparison of the functional-symptom pattern between pre- and post-operative, verified by the scores Oswestry Disability Index (ODI), Visual Analogue Scale (VAS) and EuroQol (EQ-5D);
   * the safety of the medical device, through the impact of any adverse events, complications, unexpected reactions, accidents.
4. STUDY DESIGN

4.1. Study characteristics This collection of clinical data is set up as post-market pilot study. It will be included in the study all consecutive patients who require spinal fusion surgery, in accordance with the inclusion and exclusion criteria as voluntary and after signing the informed consent. Patients will be treated and followed postoperatively according to normal clinical practice, surgical and therapeutic in place at the Rizzoli Orthopaedic Institute of Bologna.

The total duration of data collection is 36 months:

* the stage of patient enrollment is 18 months from the date of approval of the study by the Ethics Committee of the center;
* the phase of post-operative monitoring is 18 months, with planned at 6, 12 and 18 months follow-up (± 15 days before scheduled date).

In relation to the literature up to now produced, it is considered advisable to provide a post-operative control at 18 months since the chemical composition and biomimetic hydroxyapatite-magnesium shows remodeling and resorption, in a physiologically time comprised between 6 and 18 months, as well as for other reported in Section 4.

18 months is therefore the appropriate follow up to verify the medium term biomaterial behavior.

All data will be collected in a systematic, timely and uniform in a specific report form (SRD) paper.

4.2. Treatment directions Patients will be treated for degenerative diseases of the spine, such as lumbar stenosis, spondylolysis and spondylolisthesis, degenerative disc disease.

The fusion technique used will be the posterolateral arthrodesis, of one or more vertebral levels included in the lumbosacral (L1-S1), obtained by means of screws and bars, together with a preparation of the transverse processes treated with bone substitute in order to Sintlife obtain new bone formation and then spinal fusion. It also provided the ability to associate interbody posterolateral arthrodesis with the use of cage.

4.3. Visits plan During each visit (pre-operative, intra-operative, post-operative and follow-up) will be the responsibility of the surgeon to fill in the specific section in gathering data of every patient card.

The activities for each visit will be carried out as described below and as shown in the flow chart of visits (paragraph 2):

* preoperative examination (pre-op) - signing the informed consent, assessment of the criteria for inclusion - exclusion, recording demographic data and medical history, the SEA assessment and ODI;
* intervention - surgical report, TC, reports of potential adverse events intraoperative or immediate postoperative;
* follow-up visit at 6 months after surgery - report of any adverse events, the SEA assessment, ODI, EQ-5D;
* follow-up visit at 12 months after surgery - report of any adverse events, the SEA assessment, ODI, EQ-5D, TC;
* follow-up visit at 18 months after surgery - report of any adverse events, the SEA assessment, ODI, EQ-5D, TC.

ELIGIBILITY:
Inclusion Criteria:

Patients who have provided consent to the processing of personal data;

* Patients over the age of 18;
* Patients who require posterolateral fusion of lumbosacral tract (L1- S1);
* Patients suffering from traumatic and degenerative diseases of the spine, such as lumbar stenosis, spondylolysis and spondylolisthesis, degenerative disc disease;
* Patients who agree to participate in the program of visits required by the Protocol.

Exclusion Criteria:

Patients affected by:

* systemic or localized infection
* inflammatory or autoimmune disease
* hypercalcemia
* coagulation disorders
* metabolic disorders
* insulin dependent diabetes
* alterations or complications of thyroid function
* allergy to calcium phosphate
* declared allergies to medications and / or medical device
* tumor diseases and / or infectious diseases of the spine
* active neoplasia
* Patients who abuse of alcohol or drugs
* Patients in the alleged pregnancy or confirmed
* Patients on medication that causes abnormal bone regeneration (eg chemotherapy)
* Already operated patients (revision surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Spinal fusion | 18 months
  Brantigan fusion score to evaluate 5 levels of fusion

SECONDARY OUTCOMES:
Back pain assessed by VAS (Visual Analog Scale) | Change from baseline at 6, 12, 18 months
  Patient self-administered questionnaire to evaluate VAS pain score. VAS is a pain scale ranging from 0 to 10 points (where 0 is the minimum value and 10 is the maximum value). A decrease in VAS score is expected at follow up.
Functional activity assessed by ODI (Oswestry Disability Index) | Change from baseline at 6, 12, 18 months
  Patient self-administered questionnaire to evaluate the disability ODI score. ODI score is indicated as percentage ranging from 0% to 100%, where 0 corresponds to completely normal functional ability. A decrease in ODI score is expected at follow up.
Quality of life assessed by EQ-5D (Euro-QoL5D) | Change from baseline at 6, 12, 18 months
  Patient self-administered questionnaire to evaluate the quality of life (EQ5-D). EQ5-D score range from 0 to 100 points, where 0 is the minimum value and 100 is the maximum value. An increase in EQ5-D score is expected at follow up.
Adverse events | 18 months
  Evaluation of early and late adverse events emerging after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Barbanti Brodano, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdullah KG, Steinmetz MP, Benzel EC, Mroz TE. The state of lumbar fusion extenders. Spine (Phila Pa 1976). 2011 Sep 15;36(20):E1328-34. doi: 10.1097/BRS.0b013e318209952b. PMID 21358468
- [Background] Alsaleh KA, Tougas CA, Roffey DM, Wai EK. Osteoconductive bone graft extenders in posterolateral thoracolumbar spinal fusion: a systematic review. Spine (Phila Pa 1976). 2012 Jul 15;37(16):E993-1000. doi: 10.1097/BRS.0b013e3182518859. PMID 22414999
- [Background] Barbanti Brodano G, Griffoni C, Zanotti B, Gasbarrini A, Bandiera S, Ghermandi R, Boriani S. A post-market surveillance analysis of the safety of hydroxyapatite-derived products as bone graft extenders or substitutes for spine fusion. Eur Rev Med Pharmacol Sci. 2015 Oct;19(19):3548-55. PMID 26502842
- [Background] Brodano GB, Giavaresi G, Lolli F, Salamanna F, Parrilli A, Martini L, Griffoni C, Greggi T, Arcangeli E, Pressato D, Boriani S, Fini M. Hydroxyapatite-Based Biomaterials Versus Autologous Bone Graft in Spinal Fusion: An In Vivo Animal Study. Spine (Phila Pa 1976). 2014 May 15;39(11):E661-E668. doi: 10.1097/BRS.0000000000000311. PMID 24718060
- [Background] Carragee EJ, Hurwitz EL, Weiner BK. A critical review of recombinant human bone morphogenetic protein-2 trials in spinal surgery: emerging safety concerns and lessons learned. Spine J. 2011 Jun;11(6):471-91. doi: 10.1016/j.spinee.2011.04.023. PMID 21729796
- [Background] Dai LY, Jiang LS. Single-level instrumented posterolateral fusion of lumbar spine with beta-tricalcium phosphate versus autograft: a prospective, randomized study with 3-year follow-up. Spine (Phila Pa 1976). 2008 May 20;33(12):1299-304. doi: 10.1097/BRS.0b013e3181732a8e. PMID 18496340
- [Background] Dimar JR 2nd, Glassman SD, Burkus JK, Pryor PW, Hardacker JW, Carreon LY. Two-year fusion and clinical outcomes in 224 patients treated with a single-level instrumented posterolateral fusion with iliac crest bone graft. Spine J. 2009 Nov;9(11):880-5. doi: 10.1016/j.spinee.2009.03.013. Epub 2009 May 17. PMID 19447682
- [Background] Fischer CR, Cassilly R, Cantor W, Edusei E, Hammouri Q, Errico T. A systematic review of comparative studies on bone graft alternatives for common spine fusion procedures. Eur Spine J. 2013 Jun;22(6):1423-35. doi: 10.1007/s00586-013-2718-4. Epub 2013 Feb 26. PMID 23440339
- [Background] Gao C, Deng Y, Feng P, Mao Z, Li P, Yang B, Deng J, Cao Y, Shuai C, Peng S. Current progress in bioactive ceramic scaffolds for bone repair and regeneration. Int J Mol Sci. 2014 Mar 18;15(3):4714-32. doi: 10.3390/ijms15034714. PMID 24646912
- [Background] Gruskay JA, Basques BA, Bohl DD, Webb ML, Grauer JN. Short-term adverse events, length of stay, and readmission after iliac crest bone graft for spinal fusion. Spine (Phila Pa 1976). 2014 Sep 15;39(20):1718-24. doi: 10.1097/BRS.0000000000000476. PMID 24979140
- [Background] Gupta A, Kukkar N, Sharif K, Main BJ, Albers CE, El-Amin Iii SF. Bone graft substitutes for spine fusion: A brief review. World J Orthop. 2015 Jul 18;6(6):449-56. doi: 10.5312/wjo.v6.i6.449. eCollection 2015 Jul 18. PMID 26191491
- [Background] Hsu WK, Nickoli MS, Wang JC, Lieberman JR, An HS, Yoon ST, Youssef JA, Brodke DS, McCullough CM. Improving the clinical evidence of bone graft substitute technology in lumbar spine surgery. Global Spine J. 2012 Dec;2(4):239-48. doi: 10.1055/s-0032-1315454. Epub 2012 Oct 9. PMID 24353975
- [Background] Kaiser MG, Groff MW, Watters WC 3rd, Ghogawala Z, Mummaneni PV, Dailey AT, Choudhri TF, Eck JC, Sharan A, Wang JC, Dhall SS, Resnick DK. Guideline update for the performance of fusion procedures for degenerative disease of the lumbar spine. Part 16: bone graft extenders and substitutes as an adjunct for lumbar fusion. J Neurosurg Spine. 2014 Jul;21(1):106-32. doi: 10.3171/2014.4.SPINE14325. PMID 24980593
- [Background] Kannan A, Dodwad SN, Hsu WK. Biologics in spine arthrodesis. J Spinal Disord Tech. 2015 Jun;28(5):163-70. doi: 10.1097/BSD.0000000000000281. PMID 25978141
- [Background] Kho VK, Chen WC. Posterolateral fusion using laminectomy bone chips in the treatment of lumbar spondylolisthesis. Int Orthop. 2008 Feb;32(1):115-9. doi: 10.1007/s00264-006-0274-9. Epub 2006 Dec 19. PMID 17180686
- [Background] Kim DH, Rhim R, Li L, Martha J, Swaim BH, Banco RJ, Jenis LG, Tromanhauser SG. Prospective study of iliac crest bone graft harvest site pain and morbidity. Spine J. 2009 Nov;9(11):886-92. doi: 10.1016/j.spinee.2009.05.006. Epub 2009 Jun 18. PMID 19540168
- [Background] Korovessis P, Koureas G, Zacharatos S, Papazisis Z, Lambiris E. Correlative radiological, self-assessment and clinical analysis of evolution in instrumented dorsal and lateral fusion for degenerative lumbar spine disease. Autograft versus coralline hydroxyapatite. Eur Spine J. 2005 Sep;14(7):630-8. doi: 10.1007/s00586-004-0855-5. Epub 2005 Mar 24. PMID 15789231
- [Background] Lee JH, Hwang CJ, Song BW, Koo KH, Chang BS, Lee CK. A prospective consecutive study of instrumented posterolateral lumbar fusion using synthetic hydroxyapatite (Bongros-HA) as a bone graft extender. J Biomed Mater Res A. 2009 Sep 1;90(3):804-10. doi: 10.1002/jbm.a.32113. PMID 18615472
- [Background] Ludwig SC, Kowalski JM, Boden SD. Osteoinductive bone graft substitutes. Eur Spine J. 2000 Feb;9 Suppl 1(Suppl 1):S119-25. doi: 10.1007/pl00008317. PMID 10766068
- [Background] Manfrini M, Di Bona C, Canella A, Lucarelli E, Pellati A, D'Agostino A, Barbanti-Brodano G, Tognon M. Mesenchymal stem cells from patients to assay bone graft substitutes. J Cell Physiol. 2013 Jun;228(6):1229-37. doi: 10.1002/jcp.24276. PMID 23129455
- [Background] Miyazaki M, Tsumura H, Wang JC, Alanay A. An update on bone substitutes for spinal fusion. Eur Spine J. 2009 Jun;18(6):783-99. doi: 10.1007/s00586-009-0924-x. Epub 2009 Mar 12. PMID 19280232
- [Background] Nickoli MS, Hsu WK. Ceramic-based bone grafts as a bone grafts extender for lumbar spine arthrodesis: a systematic review. Global Spine J. 2014 Aug;4(3):211-6. doi: 10.1055/s-0034-1378141. Epub 2014 Jun 9. PMID 25083364
- [Background] Park JJ, Hershman SH, Kim YH. Updates in the use of bone grafts in the lumbar spine. Bull Hosp Jt Dis (2013). 2013;71(1):39-48. PMID 24032582
- [Background] Rajaee SS, Bae HW, Kanim LE, Delamarter RB. Spinal fusion in the United States: analysis of trends from 1998 to 2008. Spine (Phila Pa 1976). 2012 Jan 1;37(1):67-76. doi: 10.1097/BRS.0b013e31820cccfb. PMID 21311399
- [Background] Yoshihara H, Yoneoka D. National trends in the surgical treatment for lumbar degenerative disc disease: United States, 2000 to 2009. Spine J. 2015 Feb 1;15(2):265-71. doi: 10.1016/j.spinee.2014.09.026. Epub 2014 Oct 2. PMID 25281920
- [Background] Zhou H, Lee J. Nanoscale hydroxyapatite particles for bone tissue engineering. Acta Biomater. 2011 Jul;7(7):2769-81. doi: 10.1016/j.actbio.2011.03.019. Epub 2011 Apr 1. PMID 21440094